CLINICAL TRIAL: NCT02315963
Title: Feedback and Rewards to Increase Motivation for Therapy in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cereneo AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KFSP Feedback Study
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention group (No Intervention): Patients in stroke rehabilitation receiving standard therapy
- Intervention group (Active Comparator): Patients in stroke rehabilitation receiving standard therapy plus performance feedback
  Interventions: Other: Performance Feedback

INTERVENTIONS:
Other: Performance Feedback — Performance Feedback regarding the patients efforts and accomplishments during the patients stay in the rehabilitation clinic, an expected average of 6 weeks. The data available about the patients progress will be analysed and processed to create a visual illustration shown to the patient on a daily bases.
  Arms: Intervention group

SUMMARY:
High motivation is a predictor for good therapy results in physical therapy [Grahn 2000]. The investigator want to show that it is possible to increase patients motivation for stroke rehabilitation by providing them objective performance feedback about the patients therapy progress.

DETAILED DESCRIPTION:
High motivation is a predictor for good therapy results in physical therapy [Grahn 2000]. Additional focus on motivation and rewards has fallen on the topic of stroke rehabilitation since it was shown in an animal model that the brain centers involved with motivation and rewards are crucial to motor learning [Hosp 2011].

The investigators goal is to target the overall motivation for therapy. During the guided therapy sessions the therapists will be the main motivators and the investigators do not want to interfere with that. But the amount of guided therapy sessions is often limited due to economical reason rather than therapeutic ones. Therefore patients are encouraged to do training on their own if possible and to be active during the patients stay in the rehabilitation clinic. The investigators target the patients motivation to train by themselves and be active but also the patients attitude towards the guided therapies. It is known that performance feedback can improve motivation [Harackiewicz 1979]. Therefore the investigators want to use the data about therapy progress to produce feedback for patients visualizing the patients progress and efforts during the patients stay in the clinic.

The investigators will compare patients who receive normal therapy to patients who receive normal therapy plus performance feedback regarding a variety of motivation measures.

ELIGIBILITY:
Inclusion Criteria:

* First time Inpatient at the Cereneo rehabilitation clinic

Exclusion Criteria:

* Rey-Figur Kopie <= 25 AND Rechnerisches Denken WIE <=5
* Becks Depression Inventar (BDI) > 17
* Major aphasia preventing understanding of study materials (according to the treating physician).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Motivation | Weekly for the duration of the participants stay at the hospital an expected average of 6 weeks
  Weekly: Intrinsic Motivation Inventory Questionnaire
Motivation | After each therapy session for the duration of the participants stay at the hospital an expected average of 6 weeks
  Motivation rating of patients regarding the foregoing therapy session by therapists
Motivation | Continuous for the duration of the participants stay at the hospital an expected average of 6 weeks
  Time patient spends on self administered training
Motivation | Continuousfor the duration of the participants stay at the hospital an expected average of 6 weeks
  Amount of activities (walking, stair climbing) during free time

SECONDARY OUTCOMES:
Clinical scores (e.g. Fugl-Meyer Score) | When decided by therapists for the duration of the participants stay at the hospital an expected average of 6 weeks
  Standard quality assessments of the study site (rehabilitation clinic)

CONTACTS AND LOCATIONS:
Locations (1):
- Cereneo, Center For Rehabilitation and Neurology, Vitznau, Canton of Lucerne, Switzerland

REFERENCES:
- [Background] Grahn B, Ekdahl C, Borgquist L. Motivation as a predictor of changes in quality of life and working ability in multidisciplinary rehabilitation. A two-year follow-up of a prospective controlled study in patients with prolonged musculoskeletal disorders. Disabil Rehabil. 2000 Oct 15;22(15):639-54. doi: 10.1080/096382800445443. PMID 11087060
- [Background] Hosp JA, Pekanovic A, Rioult-Pedotti MS, Luft AR. Dopaminergic projections from midbrain to primary motor cortex mediate motor skill learning. J Neurosci. 2011 Feb 16;31(7):2481-7. doi: 10.1523/JNEUROSCI.5411-10.2011. PMID 21325515
- [Background] Harackiewicz, Judith M. The effects of reward contingency and performance feedback on intrinsic motivation. Journal of Personality and Social Psychology, Vol 37(8), Aug 1979, 1352-1363.